CLINICAL TRIAL: NCT01658826
Title: A Double-blind, Double Dummy, Randomized Crossover Trial to Compare the Effect of "AIC316 (Pritelivir)" 100 mg Once Daily Versus Valacyclovir 500 mg Once Daily on Genital HSV Shedding in HSV-2 Seropositive Adults.
Brief Title: Safety and Efficacy Comparator Trial of a New Drug Against Genital Herpes
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: AiCuris Anti-infective Cures AG (Industry)
Collaborators: Medpace, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: AIC316-01-II-02
Record Dates: First submitted 2012-08-03; First posted 2012-08-07 (Estimated); Results first posted 2023-04-21 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Genital Herpes
Keywords: AIC316; Viral shedding
MeSH Terms: conditions — Herpes Genitalis | interventions — pritelivir; Valacyclovir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- AIC316, Then Valacyclovir (Experimental): Participants first received AIC316 100 mg once daily for 28 days. After a washout period of 28 days, they then received Valacyclovir 500 mg once daily for 28 days.
  Interventions: Drug: AIC316; Drug: Valacyclovir
- Valacyclovir, Then AIC316 (Active Comparator): Participants first received Valacyclovir 500 mg once daily for 28 days. After a washout period of 28 days, they then received AIC316 100 mg once daily for 28 days.
  Interventions: Drug: AIC316; Drug: Valacyclovir

INTERVENTIONS:
Drug: AIC316 — 100 mg oral administration
Drug: Valacyclovir — 500 mg oral administration

SUMMARY:
The aim of the study is to evaluate the safety and efficacy of "AIC316 (pritelivir)" 100 mg once daily compared to valacyclovir 500 mg once daily for the prevention of HSV-2 genital shedding.

DETAILED DESCRIPTION:
Enrolled patients with Mucocutaneous genital HSV, will be randomized to receive either AIC326 or Valacyclovir first and then will be crossed over to receive the opposite Intervention. The study will consist of two treatment periods of 28 days separated by a washout period of 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Adult, immunocompetent men and women in good health of any ethnic group
* Seropositive for Herpes Simplex Virus Type 2 (HSV-2)
* History of recurrent episodes (>=4 to <=9) of genital herpes for at least 12 months and willingness to obtain 4 swabs per day.

Exclusion Criteria:

* Present episode of genital herpes at time of randomization
* Clinically relevant acute or chronic infections (excluding HSV-2)
* Known intolerance to valacyclovir, acyclovir, or any component of the formulation
* Documented HSV resistance to acyclovir, valacyclovir, famciclovir or penciclovir

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2012-10; Primary Completion 2013-05 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Indiana University School of Medicine, IU Infectious Diseases Research, Indianapolis, Indiana
  - Westover Heights Clinic, Portland, Oregon
  - University of Texas Health Science Centre, Center for Clincial Studies, Houston, Texas
  - University of Washington, Virology Research Clinic, Seattle, Washington

REFERENCES:
- [Derived] Wald A, Timmler B, Magaret A, Warren T, Tyring S, Johnston C, Fife K, Selke S, Huang ML, Stobernack HP, Zimmermann H, Corey L, Birkmann A, Ruebsamen-Schaeff H. Effect of Pritelivir Compared With Valacyclovir on Genital HSV-2 Shedding in Patients With Frequent Recurrences: A Randomized Clinical Trial. JAMA. 2016 Dec 20;316(23):2495-2503. doi: 10.1001/jama.2016.18189. PMID 27997653

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 150 subjects were screened, 59 were screen failures (did not meet study eligibility requirements: 35, withdrawal of Consent 1, Lost to Follow-up 1, Other 22). 91 subjects were randomized.
Period: Period 1: First Intervention (28 Days)
Arm/Group | AIC316, Then Valacyclovir | Valacyclovir, Then AIC316
Started | 45 | 46
Completed | 38 | 36
Not Completed | 7 | 10
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Adverse Event | 1 | 2
Not completed — Termination of the Study by the Investigator or Sponsor | 5 | 6
Not completed — Protocol Violation | 0 | 1
Not completed — Patient was non-compliant with study medication, swabbing and maintaining diary | 0 | 1
Period: Washout Period: 28 Days
Arm/Group | AIC316, Then Valacyclovir | Valacyclovir, Then AIC316
Started | 38 | 36
Completed | 32 | 32
Not Completed | 6 | 4
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Termination of the Study by the Investigator or Sponsor | 5 | 3
Period: Period 2: Second Intervention (28 Days)
Arm/Group | AIC316, Then Valacyclovir | Valacyclovir, Then AIC316
Started | 32 | 32
Completed | 29 | 27
Not Completed | 3 | 5
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Termination of the Study by the Investigator or Sponsor | 3 | 4

BASELINE CHARACTERISTICS:
Population: All randomized subjects assign to a treatment sequence.
Groups:
- Total: Total of all reporting groups
Arm/Group | AIC316, Then Valacyclovir | Valacyclovir, Then AIC316 | Total
Number analyzed (Participants) | 45 | 46 | 91
Age, Continuous [Mean (Standard Deviation); unit: Years] | 45.2 (13.22) | 45.5 (11.4) | 45.4 (12.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 29 | 57
  Male | 17 | 17 | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 7 | 14
  Not Hispanic or Latino | 38 | 39 | 77
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 7 | 9 | 16
  White | 37 | 29 | 66
  More than one race | 1 | 5 | 6
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Within-subject Genital HSV Mucocutaneous Shedding Rate
Description: Subjects were assessed for within-subject genital HSV mucocutaneous shedding rate, as calculated by the number of HSV-positive swabs per subject relative to the total number of swabs collected per subject. The swab test detects the presence of herpes virus DNA. A swab was regarded as positive for HSV-DNA if at least 3 HSV genome copies were detected by quantitative PCR per reaction (equaling 150 copies per mL of swab collection medium). When multiple swabs were available from the same time point (e.g., genital and lesional swab), the swab with the highest copy number was retained for computation of the shedding rate.
Time Frame: 28 days
Population: All subjects who received at least one dose of trial medication and provided at least 1 analyzable genital-perianal swab (not including the training swab) during the treatment period were included in the efficacy analysis (Full Analysis Set).
Measure: Mean (Standard Deviation); unit: percentage of positive swaps per subject
Groups:
- AIC316: Participants who received AIC316 100 mg once daily in either the first 28 days or last 28 days of the study.
- Valacyclovir: Participants who received Valacyclovir 500 mg once daily in either the first 28 days or last 28 days of the study.
Arm/Group | AIC316 | Valacyclovir
Number analyzed (Participants) | 76 | 76
percentage of positive swaps per subject | 2.3 (5.2) | 4.9 (10.8)
Statistical Analysis 1: Comparison: AIC316 vs Valacyclovir; Test type: Superiority; p < 0.0001, non-linear mixed effects model; Risk Ratio (RR) = 0.43, 95% CI 2-sided [0.30 to 0.63]

2. Primary Outcome: Overall Shedding Rate
Description: Subjects were assessed for overall shedding rate as the total number of HSV-positive swabs per treatment group divided by the number of swabs collected per treatment group.
Time Frame: 28 days
Population: Full Analysis Set - defined as all randomized subjects who took trial medication at least once and provided at least 1 analyzable genital-perianal swab (not including the training swab) during the treatment period.
Measure: Number; unit: percentage of positive swabs
Arm/Group | AIC316 | Valacyclovir
Number analyzed (Participants) | 76 | 76
percentage of positive swabs | 2.4 | 5.2

ADVERSE EVENTS:
Time Frame: 28 days for each intervention
Description: AE reporting is based on the safety set versus the full analysis set
Arm/Group | AIC316 | Valacyclovir
All-Cause Mortality (participants affected / at risk) | 0/77 | 0/78
Serious Adverse Events (participants affected / at risk) | 0/77 | 0/78
Other Adverse Events (participants affected / at risk) | 48/77 | 54/78
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AIC316 (N=77) | Valacyclovir (N=78)
Upper respiratory tract infection (Infections and infestations) | 11 | 8
Vulvovaginal mycotic infection (Infections and infestations) | 3 | 3
Tooth infection (Infections and infestations) | 2 | 1
Vaginitis bacteria (Infections and infestations) | 1 | 3
Gastroenteritis viral (Infections and infestations) | 0 | 2
Sinusitis (Infections and infestations) | 2 | 0
Headache (Nervous system disorders) | 12 | 14
Dizziness (Nervous system disorders) | 3 | 3
Dysgeusia (Nervous system disorders) | 0 | 4
Nausea (Gastrointestinal disorders) | 3 | 4
Diarrhea (Gastrointestinal disorders) | 4 | 2
Hemorrhoids (Gastrointestinal disorders) | 1 | 3
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 3
Dry Mouth (Gastrointestinal disorders) | 0 | 2
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 2 | 1
Vomiting (Gastrointestinal disorders) | 0 | 2
Dry Skin (Skin and subcutaneous tissue disorders) | 2 | 2
Erythema (Skin and subcutaneous tissue disorders) | 1 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0
Fatigue (General disorders) | 3 | 5
Chills (General disorders) | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Anxiety (Psychiatric disorders) | 2 | 3
Insomnia (Psychiatric disorders) | 1 | 2
Vulvovaginal pruritus (Reproductive system and breast disorders) | 2 | 1
Contusion (Injury, poisoning and procedural complications) | 2 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 2
Flushing (Vascular disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes